CLINICAL TRIAL: NCT03512769
Title: The Restful Jaw Device: A New Way to Support and Protect the Jaw During Third Molar Extractions; Feasibility
Brief Title: Feasibility Testing of a New Way to Support the Jaw During 3rd Molar Extractions
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2854
Record Dates: First submitted 2018-03-27; First posted 2018-05-01 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Impacted Third Molar Tooth; Temporomandibular Joint Dysfunction Syndrome
Keywords: jaw support device, third molars, wisdom teeth, partially erupted or impacted
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome; Tooth, Impacted

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Restful Jaw Device — The Restful Jaw device is used to support the jaw during dental procedures including surgical removal of 3rd molars (wisdom teeth) with sedation. The device is designed to counter the downward forces placed on the mandible by clinicians during dental procedures and prevent jaw hyperextension (opening too wide) while providing a secure, stable jaw position. When 3rd molar teeth are surgically removed with sedation, a dental assistant stands behind the dental chair and supports the patient's jaw with both hands under the patient's jaw. If needed, the dental assistant also holds the jaw in a slightly forward position to maintain an open airway. This device replicates the dental assistant in holding the jaw during dental procedures.

SUMMARY:
Cross sectional observational study to assess the feasibility of using the functional prototype of the restful jaw support device to support the jaw when extracting mandibular 3rd molars using moderate/deep sedation. An additional meeting(s) will occur, after the oral and maxillofacial surgeons (OMS) have completed all treatment procedures utilizing the device and surveys are completed, to provide feedback on how the device performed.

DETAILED DESCRIPTION:
Cross sectional observational study assesses the feasibility of OMS and dental assistants using the jaw support device during mandibular 3rd molar extractions with moderate/deep sedation.

Patients presenting for surgical removal of 3rd molars will be invited to participate in the study at the time of their oral surgery consult. The OMS will determine if the patient meets eligibility criteria, explain the study and invite them to participate. At the time of 3rd molar removal, the OMS and their dental assistants will follow their standard procedures for obtaining consent from patients for 3rd molar removal with moderate/deep sedation. In addition, they will confirm the patient's interest to participate in the study, ask if they have any questions and obtain consent. A dental assistant will place the jaw support device and recheck the jaw support tightening mechanism once the positioning is comfortable for the patient. The dental assistant will recheck the jaw support tightening mechanism before the procedure begins.

The OMS will use their standard protocol for removal of the teeth. The only change will be that a dental assistant who typically stands behind the dental chair and supports the mandible with their hands and moves the jaw as indicated by the OMS will instead place and secure the device to support the jaw. A dental assistant standing behind the chair will be present at all times to readjust the device position as needed or remove the device as indicated. The default in the case of device malfunction is for the device to fall away from the patient and the dental assistant will be immediately available to take over supporting the patient's jaw with their hands, which is one of their standard responsibilities when the device is not used.

Both the OMS and any dental assistant(s) assisting in the procedure(s), when the device is utilized, will each complete a survey about their experience with the jaw support device once they have completed surgical removal with moderate/deep sedation of mandibular 3rd molars in 4 patients.

An additional meeting(s) will occur, after the OMS have completed all treatment procedures utilizing the device and surveys are completed, to provide feedback on how the device performed. This information will inform Phase II of this study, a randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 to 24 years of age.
* Requires surgical removal of bilateral mandibular 3rd molars (concurrent maxillary 3rd molar extractions allowed).
* Will consent to have 3rd molar surgical removal with the device supporting the mandible.
* Indication for moderate/deep sedation and medically able to tolerate sedation.
* American Society of Anesthesiologists (ASA) Physical Status Category I (healthy patient) and Category II (patients with mild systemic disease).

Exclusion Criteria:

• Any condition or situation that the surgeon feels would prevent the patient from participating in the study.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients that present to the participating oral and maxillofacial surgeons' office for mandibular 3rd molar surgical removal with moderate/deep sedation
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
The feasibility will be assessed by query of the surgeons utilizing the device (questionnaire). This will be done after 4 patient experiences in conjunction with surgical procedure. | 3-6 months
  Surgeons satisfaction with utilization of the device.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman JW. The prophylactic extraction of third molars: a public health hazard. Am J Public Health. 2007 Sep;97(9):1554-9. doi: 10.2105/AJPH.2006.100271. Epub 2007 Jul 31. PMID 17666691
- [Background] Huang GJ, Rue TC. Third-molar extraction as a risk factor for temporomandibular disorder. J Am Dent Assoc. 2006 Nov;137(11):1547-54. doi: 10.14219/jada.archive.2006.0090. PMID 17082281
- [Background] Huang GJ, Cunha-Cruz J, Rothen M, Spiekerman C, Drangsholt M, Anderson L, Roset GA. A prospective study of clinical outcomes related to third molar removal or retention. Am J Public Health. 2014 Apr;104(4):728-34. doi: 10.2105/AJPH.2013.301649. Epub 2014 Feb 13. PMID 24524521
- [Background] Huang GJ, Drangsholt MT, Rue TC, Cruikshank DC, Hobson KA. Age and third molar extraction as risk factors for temporomandibular disorder. J Dent Res. 2008 Mar;87(3):283-7. doi: 10.1177/154405910808700313. PMID 18296615
- [Background] Huang GJ, LeResche L, Critchlow CW, Martin MD, Drangsholt MT. Risk factors for diagnostic subgroups of painful temporomandibular disorders (TMD). J Dent Res. 2002 Apr;81(4):284-8. doi: 10.1177/154405910208100412. PMID 12097315
- [Background] Juhl GI, Jensen TS, Norholt SE, Svensson P. Incidence of symptoms and signs of TMD following third molar surgery: a controlled, prospective study. J Oral Rehabil. 2009 Mar;36(3):199-209. doi: 10.1111/j.1365-2842.2008.01925.x. PMID 19207447
- [Background] Akhter R, Hassan NM, Ohkubo R, Tsukazaki T, Aida J, Morita M. The relationship between jaw injury, third molar removal, and orthodontic treatment and TMD symptoms in university students in Japan. J Orofac Pain. 2008 Winter;22(1):50-6. PMID 18351034
- [Background] Velly AM, Gornitsky M, Philippe P. Contributing factors to chronic myofascial pain: a case-control study. Pain. 2003 Aug;104(3):491-499. doi: 10.1016/S0304-3959(03)00074-5. PMID 12927621
- [Background] Okeson JP. Bell's orofacial pains: The clinical management of orofacial pain, sixth edition. Vol 6. Illinois: Quintessence Publishing; 2005.
- [Background] Pullinger AG, Monteiro AA. History factors associated with symptoms of temporomandibular disorders. J Oral Rehabil. 1988 Mar;15(2):117-24. doi: 10.1111/j.1365-2842.1988.tb00760.x. PMID 3163728
- [Background] LeResche L, Mancl LA, Drangsholt MT, Huang G, Von Korff M. Predictors of onset of facial pain and temporomandibular disorders in early adolescence. Pain. 2007 Jun;129(3):269-278. doi: 10.1016/j.pain.2006.10.012. Epub 2006 Nov 28. PMID 17134830
- [Background] Plesh O, Gansky SA, Curtis DA, Pogrel MA. The relationship between chronic facial pain and a history of trauma and surgery. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1999 Jul;88(1):16-21. doi: 10.1016/s1079-2104(99)70187-3. PMID 10442939
- [Background] Butler JH, Folke LE, Bandt CL. A descriptive survey of signs and symptoms associated with the myofascial pain-dysfunction syndrome. J Am Dent Assoc. 1975 Mar;90(3):635-9. doi: 10.14219/jada.archive.1975.0147. PMID 1054051
- [Background] Fricton JR, Kroening R, Haley D, Siegert R. Myofascial pain syndrome of the head and neck: a review of clinical characteristics of 164 patients. Oral Surg Oral Med Oral Pathol. 1985 Dec;60(6):615-23. doi: 10.1016/0030-4220(85)90364-0. PMID 3865133
- [Background] Sahebi S, Moazami F, Afsa M, Nabavi Zade MR. Effect of lengthy root canal therapy sessions on temporomandibular joint and masticatory muscles. J Dent Res Dent Clin Dent Prospects. 2010 Summer;4(3):95-7. doi: 10.5681/joddd.2010.024. Epub 2010 Sep 16. PMID 22991607
- [Background] Humphrey SP, Lindroth JE, Carlson CR. Routine dental care in patients with temporomandibular disorders. J Orofac Pain. 2002 Spring;16(2):129-34. PMID 12043519
- [Background] American Association of Oral and Maxillofacial Surgeons. Parameters of care: Clinical and practice guidelines for oral and maxillofacial surgeons. 2012. Available at http://www.mfch.cz/doc/ParCare2012Complete.pdf
- [Background] Fernandes P, Velly AM, Anderson GC. A randomized controlled clinical trial evaluating the effectiveness of an external mandibular support device during dental care for patients with temporomandibular disorders. Gen Dent. 2013 Sep-Oct;61(6):26-31. PMID 24064159
- [Background] Zucuskie T. A controlled clinical trial of the usefulness of an external mandibular support device during routine dental care. Minneapolis: University of Minnesota; 1996.